CLINICAL TRIAL: NCT03689907
Title: Assessing the Predictive Potential of Early Chimerism Analysis Following Allogeneic Stem-Cell Transplant
Brief Title: Early Chimerism Following Allogeneic Stem-Cell Transplant
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, John M. Hill, Jr., MD, Director, Allogeneic Bone Marrow Transplant Program, Dartmouth-Hitchcock Medical Center
Other Study IDs: D18125; NCI-2020-03008 (Other: NCI ID)
Record Dates: First submitted 2018-09-27; First posted 2018-10-01 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Allogeneic Stem-Cell Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Allogeneic Stem-Cell Transplant Recipients: 1. At day +14/15-post transplant - lineage-specific chimerism analysis will be performed on a peripheral blood sample drawn from the patient.
  2. At day +30-post transplant, most participants will be in the outpatient setting and would undergo chimerism evaluation as part of the standard of care for transplant patients.
  Interventions: Other: Chimerism Evaluation

INTERVENTIONS:
Other: Chimerism Evaluation — Blood collection for chimerism evaluation will be performed on days +14/15-post transplant and +30-post transplant for each study participant.

SUMMARY:
Allogeneic stem cell transplant (allo-SCT) is a common treatment for variety of blood cancers. To determine how many cells are from the donor after transplant, doctors complete a "chimerism analysis" or a test of participant cells to look at the DNA. Chimerism testing helps doctors predict graft rejection or recurrence of disease. Doctors at NCCC do chimerism testing routinely and it is usually done between 30 and 100 days after transplantation. The researchers believe that analyzing chimerism sooner than 30 days after transplant may help identify problems earlier, get patients treatment sooner, and increase the chances of a successful transplant.

The purpose of this study is to find out if doing chimerism testing earlier than the traditional approach is better for patient outcomes (about 14 days after transplantation rather than 30+ days). Information gained from this study can be used to help prevent some post-transplant complications such as graft loss, graft-versus-host disease, or even relapse for future patients.

Also, the researchers hope to learn more about chimerism testing of cells of patients with haploidentical donors (donors who are only a "half-match" - such as a parent or child of the recipient), because there have not been many chimerism analysis studies done in this population.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have been cleared by a Transplant Attending to undergo allogeneic stem cell transplant

Exclusion Criteria:

* Patients undergoing a second allogeneic stem cell transplant or beyond

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants in this study will receive an allogeneic stem-cell transplant.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Characterize early lineage-specific chimerism profiles in allogeneic stem-cell transplant recipients | 14 or 15 days post-transplant
  Our method of chimerism analysis is dependent on baseline DNA samples of pre-transplant donor and recipient, then serial assessment of polymorphic short tandem repeats (STRs) to specifically characterize the source (donor vs recipient) of DNA extracted from our patients' leukocytes at day +14/15 after allogeneic stem cell transplant. First, DNA is extracted from the buffy coat layer of an EDTA blood sample, then PCR reactions using STR markers are prepared, and the differently sized fluorescent PCR products are then assessed on a genetic analyzer. An assessment of the relative amounts of donor and recipient chimerism can then be determined from the analyzer output, based on peak height and area. The discreet leukocyte lineages are then isolated by cell separation, and DNA is isolated from these purified fractions and assessed as for whole blood.

SECONDARY OUTCOMES:
Correlate early chimersim profiles with donor chimerism | Day +30-post transplant
  Day +14/15-post transplant absolute neutrophil count and absolute lymphocyte count will be compared to the Day +30-post transplant lineage-specific chimerism profile to determine if there is a correlation between early lineage chimerism and full donor chimerism.

CONTACTS AND LOCATIONS:
Overall Officials: John M. Hill, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Farhan S, Bazydlo M, Neme K, Mikulandric N, Peres E, Janakiraman N. Chimerism in Myeloid Malignancies following Stem Cell Transplantation Using FluBu4 with and without Busulfan Pharmacokinetics versus BuCy. Adv Hematol. 2017;2017:8690416. doi: 10.1155/2017/8690416. Epub 2017 Nov 8. PMID 29250116
- [Background] Passweg JR, Baldomero H, Bader P, Bonini C, Duarte RF, Dufour C, Gennery A, Kroger N, Kuball J, Lanza F, Montoto S, Nagler A, Snowden JA, Styczynski J, Mohty M. Use of haploidentical stem cell transplantation continues to increase: the 2015 European Society for Blood and Marrow Transplant activity survey report. Bone Marrow Transplant. 2017 Jun;52(6):811-817. doi: 10.1038/bmt.2017.34. Epub 2017 Mar 13. PMID 28287639
- [Background] Parmesar K, Raj K. Haploidentical Stem Cell Transplantation in Adult Haematological Malignancies. Adv Hematol. 2016;2016:3905907. doi: 10.1155/2016/3905907. Epub 2016 May 30. PMID 27313619
- [Background] Fabricius WA, Ramanathan M. Review on Haploidentical Hematopoietic Cell Transplantation in Patients with Hematologic Malignancies. Adv Hematol. 2016;2016:5726132. doi: 10.1155/2016/5726132. Epub 2016 Feb 29. PMID 27034676
- [Background] Bashey A, Solomon SR. T-cell replete haploidentical donor transplantation using post-transplant CY: an emerging standard-of-care option for patients who lack an HLA-identical sibling donor. Bone Marrow Transplant. 2014 Aug;49(8):999-1008. doi: 10.1038/bmt.2014.62. Epub 2014 May 19. PMID 24842530
- [Background] Koreth J, Kim HT, Nikiforow S, Milford EL, Armand P, Cutler C, Glotzbecker B, Ho VT, Antin JH, Soiffer RJ, Ritz J, Alyea EP 3rd. Donor chimerism early after reduced-intensity conditioning hematopoietic stem cell transplantation predicts relapse and survival. Biol Blood Marrow Transplant. 2014 Oct;20(10):1516-21. doi: 10.1016/j.bbmt.2014.05.025. Epub 2014 Jun 4. PMID 24907627
- [Background] Reshef R, Hexner EO, Loren AW, Frey NV, Stadtmauer EA, Luger SM, Mangan JK, Gill SI, Vassilev P, Lafferty KA, Smith J, Van Deerlin VM, Mick R, Porter DL. Early donor chimerism levels predict relapse and survival after allogeneic stem cell transplantation with reduced-intensity conditioning. Biol Blood Marrow Transplant. 2014 Nov;20(11):1758-66. doi: 10.1016/j.bbmt.2014.07.003. Epub 2014 Jul 10. PMID 25016197
- [Background] Mathur, A and Malhotra, H. Haploidentical Stem Cell Transplantation: A Mini Review. J Stem Cell Res Ther 2017; 2(2): 00056.
- [Background] Mattsson J, Ringden O, Storb R. Graft failure after allogeneic hematopoietic cell transplantation. Biol Blood Marrow Transplant. 2008 Jan;14(1 Suppl 1):165-70. doi: 10.1016/j.bbmt.2007.10.025. Erratum In: Biol Blood Marrow Transplant. 2008 Nov;14(11):1317-8. PMID 18162238
- [Background] Legrand, F et al. Chimerism Analysis after Haploidentical Stem Cell Transplantation: Is It Necessary for All Patients? Blood 2016; 128: 3417.
- [Background] Hussain, A et al. Lineage-Specific Chimerism and Incidence of Graft Failure Following T-Cell Replete Haploidentical Transplantation Using Post-Transplant Cyclophosphamide in Eighty-Nine Consecutive Patients From a Single Center. Blood 2012; 120: 3030.
- [Background] Moscardo F, Sanz J, Senent L, Cantero S, de la Rubia J, Montesinos P, Planelles D, Lorenzo I, Cervera J, Palau J, Sanz MA, Sanz GF. Impact of hematopoietic chimerism at day +14 on engraftment after unrelated donor umbilical cord blood transplantation for hematologic malignancies. Haematologica. 2009 Jun;94(6):827-32. doi: 10.3324/haematol.2008.000935. PMID 19483157
- [Background] Miura Y, Tanaka J, Toubai T, Tsutsumi Y, Kato N, Hirate D, Kaji M, Sugita J, Shigematsu A, Iwao N, Ota S, Masauzi N, Fukuhara T, Kasai M, Asaka M, Imamura M. Analysis of donor-type chimerism in lineage-specific cell populations after allogeneic myeloablative and non-myeloablative stem cell transplantation. Bone Marrow Transplant. 2006 May;37(9):837-43. doi: 10.1038/sj.bmt.1705352. PMID 16547484
- [Background] Breuer S, Preuner S, Fritsch G, Daxberger H, Koenig M, Poetschger U, Lawitschka A, Peters C, Mann G, Lion T, Matthes-Martin S. Early recipient chimerism testing in the T- and NK-cell lineages for risk assessment of graft rejection in pediatric patients undergoing allogeneic stem cell transplantation. Leukemia. 2012 Mar;26(3):509-19. doi: 10.1038/leu.2011.244. Epub 2011 Sep 16. PMID 21926962
- [Background] Choi, YB et al. Does Day 14 Peripheral Blood Chimerism after Allogeneic Hematopoietic Stem Cell Transplantation Predict Treatment Failure in Children with Non-Malignant Disease? BBMT 2016; 22: S310.
- [Background] Antin JH, Childs R, Filipovich AH, Giralt S, Mackinnon S, Spitzer T, Weisdorf D. Establishment of complete and mixed donor chimerism after allogeneic lymphohematopoietic transplantation: recommendations from a workshop at the 2001 Tandem Meetings of the International Bone Marrow Transplant Registry and the American Society of Blood and Marrow Transplantation. Biol Blood Marrow Transplant. 2001;7(9):473-85. doi: 10.1053/bbmt.2001.v7.pm11669214.
- [Background] Huisman C, de Weger RA, de Vries L, Tilanus MG, Verdonck LF. Chimerism analysis within 6 months of allogeneic stem cell transplantation predicts relapse in acute myeloid leukemia. Bone Marrow Transplant. 2007 Mar;39(5):285-91. doi: 10.1038/sj.bmt.1705582. Epub 2007 Jan 29. PMID 17262061